CLINICAL TRIAL: NCT01581606
Title: Evaluation of TeleOphthalmology in Age-related Macular Degeneration (AMD) - TeleMedicine Solutions to Improve Patient Access and Quality of Vision Outcomes.
Brief Title: Evaluation of TeleOphthalmology in AMD-TeleMedicine Solutions to Improve Patient Access and Quality of Vision Outcomes
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Academic Health Science Centres (Other)
Responsible Party: Sponsor
Other Study IDs: 18045E
Record Dates: First submitted 2012-04-12; First posted 2012-04-20 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Age Related Macular Degeneration
Keywords: Age Related Macular Degeneration; Teleophthalmology; Screening; Diagnosis; Timing; Treatment
MeSH Terms: conditions — Macular Degeneration; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1R and 1T AMD Screening: Group 1 patients will be collected through all referrals to any of the physician investigators with a provisional diagnosis of possible wet AMD. Any request for clinical evaluation of a patient for presumed wet AMD will be randomized into Group 1R (Routine Screening) and Group 1T (Tele-ophthalmology screening).
- Group 2R and 2T Follow up: Group 2 patients will be collected from the patients previously treated for wet AMD within the practices of the physician investigators. All patients in whom the disease is inactive (not receiving active treatment) and who therefore require monitoring will be randomized into Group 2R (Routine Monitoring) and Group 2T (Teleophthalmology Monitoring).

SUMMARY:
Hypothesis:

The use of teleophthalmology for patient screening will result in more rapid patient access for treatment. The use of teleophthalmology to monitor patients with wet AMD post-treatment will result in maintenance of good visual outcomes combined with a reduction in patient travel and improved patients satisfaction in a cost effective manner.

Objectives :

The Evaluation of Teleophthalmology in AMD project objectives are as follows:

1. To evaluate the efficacy of teleophthalmology in screening patients referred to retina specialists for suspected wet AMD.
2. To compare the "time to treatment/retreatment" with this program with that of patient's entering the system and being followed conventionally to determine the efficacy of teleophthalmology to provide rapid entry/re-entry into treatment programs.
3. To determine the efficacy of teleophthalmology in monitoring patients with wet AMD post therapy.
4. To determine the compliance rate for monitoring wet AMD during follow-up utilizing teleophthalmology.
5. To evaluate the cost effectiveness of teleophthalmology in screening/monitoring wet AMD patients including direct costs to the OHIP system and indirect costs to the patient/caregiver.
6. To assess patient satisfaction with teleophthalmology versus standard clinical care in the monitoring of post-treatment wet AMD.
7. To evaluate teleophthalmology as a tool for communication between community based Optometrists /Ophthalmologists and Retina Specialists.

DETAILED DESCRIPTION:
For purposes of this study, two patient streams will be developed and implemented: AMD screening patients (Group 1) and post-Lucentis monitoring patients (Group 2).

Group 1 patients will be collected through all referrals to any of the physician investigators with a provisional diagnosis of possible wet AMD. Any request for clinical evaluation of a patient for presumed wet AMD will be randomized into Group 1R (Routine Screening) and Group 1T (Tele-ophthalmology screening).

In group 1R patients will receive an appointment in the current standard fashion with review and consultation within the retinal physician's office, evaluation of the need for diagnostic testing and subsequent treatment as indicated. Group 1T will undergo pre-screening at the nearest OHC. These patients will obtain full ocular evaluation by the current OTN (Ontario Telemedicine Network) ophthalmology pilot standards (visual acuity, intraocular pressure measurement, fundus photography and OCT - at a quality level established by a working group for the OTN in 2009). At the completion of the screening visit, images and data will be stored in the OHC database and notification of the visit sent to the treating center. This will trigger a formal evaluation and grading of the patient's status and determination of the need for an in person evaluation and treatment at the treating center. This formal evaluation will occur only if the teleophthalmology dataset suggests the presence of wet AMD requiring treatment or if the dataset quality is insufficient to allow accurate determination of the need to treat. In both groups following consultation, a full report for each patient will be generated which documents the patient's current macular status and suggested management strategy.

Group 2 patients will be collected from the patients previously treated for wet AMD within the practices of the physician investigators. All patients in whom the disease is inactive (not receiving active treatment) and who therefore require monitoring will be randomized into Group 2R (Routine Monitoring) and Group 2T (Teleophthalmology Monitoring).

As in group 1, patients in Group 2T will obtain a full ocular evaluation by the current OTN (Ontario Telemedicine Network) ophthalmology pilot standards, and as in group 1, this data will be analyzed to determine the need for retreatment. If necessary, the patients will be recalled to the treating center. Those who do not meet the requirements for retreatment will be booked for reassessment in two months. The two month follow up period, although longer than the "gold standard", is the routine being employed clinically at this time across the province. This is due to the current OHIP rules which cover the costs associated with OCT to a maximum of 6 per year and a desire to limit the out of pocket expenses patients incur. The follow up period of two months will be standard in both groups 2T and 2R.

Group 2R patients will be reviewed in person with evaluation in the standard fashion by obtaining visual acuity, fundus photography and OCT within the investigators clinic and will receive treatment following this consultation as needed on the date of that visit.

Data will be collected, stored, and transmitted in a secure password protected manner with appropriate encryption.

Data to be obtained will include participant age, sex, number and type of prior AMD treatments, current driving status, distance from the site of residence to the screening and treatment sites respectively. Data to answer objective 2 will be obtained by the research coordinator at study entry including duration of visual symptoms, time (in weeks) from initiation of symptoms to initial assessment visit and time (in weeks) between initial assessment and screening visit to determine treatment eligibility), time from monitoring visit to treatment, and the number of visits not requiring treatment (deemed "avoidable"). The study will included a short, post screening visit patient satisfaction questionnaire to assess the perceived patient satisfaction with the screening/monitoring process to answer objective 6. In patients who are being followed after treatment, additional demographics from the office of the vitreoretinal surgeons will be collected including baseline visual acuity, and prior treatments (in each eye and number of treatments).

Data will be collected to document patient compliance with scheduled visits, the timing of evaluations, the imaging quality/adequacy as perceived by the grading physician, recurrent disease activity and recurrence rate, and time from the assessment visits treatment if applicable. Patients will also be administered a short patient satisfaction survey regarding duration of visit, parking / facility access, perceived satisfaction with clinic or OHC visit. These questionnaires will be done at discharge from the hospital system, at the completion of the first OHC visit and at the end of 1 year of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Patients will be collected from all referrals with a provisional diagnosis of possible Wet-AMD to any of the physician investigators. These patients will subsequently be randomized into Group 1R (Routine Screening) and Group 1T (Tele-ophthalmology Screening)
* Group 2: Patients will be collected from patients previously treated at this institution for Wet-AMD within the practices of the physician investigators. All patients in whom the disease is inactive (not receiving active treatment) and who require monitoring will be randomized into Group 2R (Routine Monitoring) and Group 2T (Tele-Ophthalmology Monitoring).

Exclusion Criteria:

* Patients will be excluded if they live more than an hours driving distance from London or from one of the afore-mentioned Ocular Health Centre(s)
* Patients with a presumed diagnosis of Wet-AMD at the time of referral who have previously had diagnostic imaging performed as part of the referral will be excluded.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: Patients will be collected from all referrals with a provisional diagnosis of possible Wet-AMD to any of the physician investigators.
  Group 2: Subjects will be collected from patients previously treated at this institution for wet-AMD within the practices of the physician investigators.
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2013-04-30 (Actual); Primary Completion 2014-04-04 (Actual); Study Completion 2014-04-07 (Actual)

PRIMARY OUTCOMES:
Wait time for treatment (naive versus follow-up patients). | One month for Tele-screening evaluation in both groups.

SECONDARY OUTCOMES:
Patient satisfaction. | One month.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Sheidow, MD, FRCSC, Principal Investigator — Ivey Eye Institute, St. Joseph's Health Care, London, Ontario, Canada
Locations (1):
- Ivey Eye Institute, St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Derived] Li B, Powell AM, Hooper PL, Sheidow TG. Prospective evaluation of teleophthalmology in screening and recurrence monitoring of neovascular age-related macular degeneration: a randomized clinical trial. JAMA Ophthalmol. 2015 Mar;133(3):276-82. doi: 10.1001/jamaophthalmol.2014.5014. PMID 25473945